CLINICAL TRIAL: NCT00385684
Title: Low-Dose Opiate Therapy for Discomfort in Dementia (L-DOT)
Acronym: LDOT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: F4483-I
Record Dates: First submitted 2006-10-06; First posted 2006-10-11 (Estimated); Results first posted 2015-11-20 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Alzheimer Disease; Dementia; Dementia, Vascular; Pain
Keywords: Agitation; Alzheimer Disease; Analgesics; Dementia; Narcotics; Opioid; Pain; Palliative Care; Psychomotor; Suffering, Physical
MeSH Terms: conditions — Alzheimer Disease; Dementia; Dementia, Vascular; Pain; Psychomotor Agitation | interventions — oxycodone-acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A1: hydrocodone/APAP w placebo PRN (Experimental): This is a fully crossed study, each participant serves as his own control. Phase A (closed label) has two arms: A1 is the experimental and A2 is the placebo comparator. Participants are randomized to either A1 for 1 week then A2 for 1 week OR A2 for 1 week then A1 for one week. A1: hydrocodone/acetaminophen 2.5/167 mg per 5 ml liquid TID, with liquid placebo available PRN. A2: liquid placebo TID with hydrocodone/acetaminophen 2.5/167 mg per 5 ml liquid PRN.
  Interventions: Drug: hydrocodone/APAP w placebo PRN
- A2: placebo w hydrocodone/APAP PRN (Placebo Comparator): This is a fully crossed study, each participant serves as his own control. Phase A: Participants are randomized to either A1 for 1 week then A2 for 1 week OR A2 for 1 week then A1 for one week. A1: hydrocodone/acetaminophen 2.5/167 mg per 5 ml liquid TID, with liquid placebo available PRN. A2: liquid placebo TID with hydrocodone/acetaminophen 2.5/167 mg per 5 ml liquid PRN.
  Interventions: Drug: placebo with hydrocodone/APAP PRN
- B: Open label hydrocodone/acetaminophen (Active Comparator): Phase B: If tolerated study medication during Phase A (i.e., the closed label, double-blind phase of the trial) then enter a six-week, open-label phase. Participants judged as responders during Phase A continue the same dose of study medication. Otherwise, moved to a higher dose (hydrocodone/acetaminophen 5/500mg TID or the most appropriate formulary alternative). Participant can also receive up to 2 PRN administrations at the same dose levels as listed above, but not to exceed 2.5g of acetaminophen.
  Interventions: Drug: hydrocodone/APAP

INTERVENTIONS:
Drug: hydrocodone/APAP w placebo PRN — Hydrocodone/acetaminophen 2.5/167 mg per 5 ml liquid three times daily (TID). With liquid placebo available PRN.
  Other Names: Lortab
  Arms: A1: hydrocodone/APAP w placebo PRN
Drug: hydrocodone/APAP — Participants judged as responders during Phase A continue the same dose of study medication (hydrocodone/acetaminophen 2.5/167 mg per 5 ml liquid TID). Otherwise, moved to a higher dose (hydrocodone/acetaminophen 5/500mg TID or the most appropriate formulary alternative). Participant can also receive up to 2 PRN administrations at the same dose levels as listed above, but not to exceed 2.5g of acetaminophen.
  Other Names: Lortab
  Arms: B: Open label hydrocodone/acetaminophen
Drug: placebo with hydrocodone/APAP PRN — Liquid placebo PRN. Also available PRN is Hydrocodone/acetaminophen 2.5/167 mg per 5 ml liquid.
  Other Names: placebo with Lortab PRN
  Arms: A2: placebo w hydrocodone/APAP PRN

SUMMARY:
The purpose of this study was to determine whether a low dose an opiate pain medication is effective for the treatment of discomfort in patients with advanced dementia. The study medication was also known as Lortab and contained both a narcotic pain medication and acetaminophen (the same pain medication as contained in Tylenol). This study was an eight-week long clinical trial for discomfort among veterans with advanced dementia who were admitted to a Nursing Home Care Unit (NHCU) at the Tuscaloosa VA Medical Center.

DETAILED DESCRIPTION:
OBJECTIVES: The primary objective of the Low-Dose Opiate Therapy for Discomfort in Dementia (L-DOT) project was to determine whether low-dose opiates are effective and well tolerated for the treatment of pain (as manifest by discomfort) in patients with advanced dementia.

RESEARCH DESIGN: This study was a two-week double-blind, double-dummy, placebo-controlled, crossover trial of low-dose hydrocodone/acetaminophen (Lortab) for discomfort among veterans with a dementia, followed by six weeks of open-label therapy for patients who tolerated treatment during the first two weeks (eight weeks total treatment on study).

METHODOLOGY: After consent, patients over age 55 with dementia residing in a nursing home care unit (or at home who receive care) at Tuscaloosa VAMC who demonstrate significant discomfort (as measured by the Pain Assessment in Advanced Dementia - PAINAD) were randomized to one of two groups, using a double-blind, double-dummy, placebo-controlled, crossover design. Patients were randomly assigned to treatment with either hydrocodone/acetaminophen 2.5mg/250mg q8hrs scheduled with placebo q8hrs PRN or placebo q8hrs scheduled with hydrocodone/acetaminophen 2.5mg/250mg q8hrs PRN. After one week's treatment, patients were crossed over to the other (opposite) regimen, for a total of two weeks of blinded treatment. Patients who tolerated treatment with hydrocodone/acetaminophen were eligible for a six-week, open-label continuation phase. The primary outcome measure was pain/discomfort. Preliminary sample size calculations indicated that 42 patients (48 patients accounting for dropouts) would be needed to be enrolled over three years to detect a difference between treatments with power of .80 and two-tailed alpha of .05.

SIGNIFICANCE: There is evidence that pain is both under recognized and undertreated in long term care settings. This study hoped to make a significant contribution to the evidence base for a common and problematic situation among veterans with advanced dementia. Advances in pain and symptom control are central to the improvement of palliative care intervention for dementia patients. Low-dose opiates are the logical next category of analgesics to consider, but have been rarely studied for this purpose in this population.

ELIGIBILITY:
Inclusion Criteria:

* 55 years of age or older;
* Must have a diagnosis of dementia;
* Advanced stage of dementia demonstrated by a score of 6 or greater on the Functional Assessment Staging (FAST) scale;
* Unable to report pain in a reliable and consistent manner;
* Have a PAINAD score of at least 2 on two consecutive assessments (separated by at least two days) OR an average PAINAD score of at least 2 on three consecutive assessments each separated by at least two days;
* The patient must have at least one medical condition associated with pain recorded on the CPRS problem list.

Exclusion Criteria:

* The existence of an effective analgesia treatment regimen;
* Pain treatment related to angina or pain judged to be related to angina;
* Current pain treatment with opiates that cannot, in the opinion of the attending physician, be discontinued without placing the patient at risk for increased pain or opiate withdrawal;
* Current pain treatment with tramadol that cannot, in the opinion of the attending physician, be discontinued;
* Presence of necessary drug therapy that is incompatible with or has potential for clinically significant drug interaction with either hydrocodone or acetaminophen;
* A history of allergy, hypersensitivity, or intolerance to either hydrocodone or acetaminophen;
* Constipation refractory to current treatment measures or a condition that would make constipation dangerous for the patient in the opinion of the attending physician;
* The presence of liver disease, hepatic encephalopathy, or clinically significant elevation of liver function tests (LFTs), as determined by the attending physician;
* The presence of renal failure, clinically significant renal insufficiency, or clinically significant elevations of serum BUN or creatinine levels, as determined by the attending physician; OR
* Evidence, based on assessment by a geriatrician, that the apparent behavioral manifestations of discomfort are better explained by another problem (e.g., fever, infection, dehydration, delirium, psychosis)

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2007-10; Primary Completion 2011-12 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Snow, PhD MS BS, Principal Investigator — VA Medical Center, Tuscaloosa
Locations (3):
- United States (3):
  - Tuscaloosa VA Medical Center, Tuscaloosa, Alabama
  - Tuscaloosa Veterans Affairs Medical Center, Tuscaloosa, Alabama
  - VA Medical Center, Tuscaloosa, Tuscaloosa, Alabama

RESULTS

PARTICIPANT FLOW:
Groups:
- A1 and Then A2 Then Phase B; A2 THEN A1 Then Phase B: This is a fully crossed study, each participant serves as his own control. Phase A: Participants are randomized to either A1 for 1 week then A2 for 1 week OR A2 for 1 week then A1 for one week. A1: hydrocodone/acetaminophen 2.5/167 mg per 5 ml liquid TID, with liquid placebo available PRN. A2: liquid placebo TID with hydrocodone/acetaminophen 2.5/167 mg per 5 ml liquid PRN.
  Phase B: If tolerated study medication during Phase A (i.e., the closed label, double-blind phase of the trial) then enter a six-week, open-label phase. Participants judged as responders during Phase A continue the same dose of study medication. Otherwise, moved to a higher dose (hydrocodone/acetaminophen 5/500mg TID or the most appropriate formulary alternative). Participant can also receive up to 2 PRN administrations at the same dose levels as listed above, but not to exceed 2.5g of acetaminophen.
Period: FIRST INTERVENTION OF PHASE A
Arm/Group | A1 and Then A2 Then Phase B | A2 THEN A1 Then Phase B
Started | 6 | 5
Completed | 5 | 5
Not Completed | 1 | 0
Not completed — Death | 1 | 0
Period: SECOND INTERVENTION OF PHASE A
Arm/Group | A1 and Then A2 Then Phase B | A2 THEN A1 Then Phase B
Started | 5 | 5
Completed | 5 | 3
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — study drug recall | 0 | 1
Period: PHASE B
Arm/Group | A1 and Then A2 Then Phase B | A2 THEN A1 Then Phase B
Started | 5 | 3
Completed | 5 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Veterans with severe dementia residing in VA nursing home.
Groups:
- ALL STUDY PARTICIPANTS: This is a fully crossed study, each participant serves as his own control. Phase A: Participants are randomized to either A1 for 1 week then A2 for 1 week OR A2 for 1 week then A1 for one week. A1: hydrocodone/acetaminophen 2.5/167 mg per 5 ml liquid TID, with liquid placebo available PRN. A2: liquid placebo TID with hydrocodone/acetaminophen 2.5/167 mg per 5 ml liquid PRN.
  Phase B: If tolerated study medication during Phase A (i.e., the closed label, double-blind phase of the trial) then enter a six-week, open-label phase. Participants judged as responders during Phase A continue the same dose of study medication. Otherwise, moved to a higher dose (hydrocodone/acetaminophen 5/500mg TID or the most appropriate formulary alternative). Participant can also receive up to 2 PRN administrations at the same dose levels as listed above, but not to exceed 2.5g of acetaminophen.
Arm/Group | ALL STUDY PARTICIPANTS
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 11

OUTCOME MEASURES:

1. Primary Outcome: Pain Assessment in Advanced Dementia (PAINAD)
Description: Pain intensity observational assessment for persons with severe dementia. Higher scores indicate more pain/discomfort. Scale range is 0-10.
Time Frame: Two (2) weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Experimental: A1; Placebo Comparator: A2: This is a fully crossed study, each participant serves as his own control. Phase A: Participants are randomized to either A1 for 1 week then A2 for 1 week OR A2 for 1 week then A1 for one week. A1: hydrocodone/acetaminophen 2.5/167 mg per 5 ml liquid TID, with liquid placebo available PRN. A2: liquid placebo TID with hydrocodone/acetaminophen 2.5/167 mg per 5 ml liquid PRN.
  Phase B: If tolerated study medication during Phase A (i.e., the closed label, double-blind phase of the trial) then enter a six-week, open-label phase. Participants judged as responders during Phase A continue the same dose of study medication. Otherwise, moved to a higher dose (hydrocodone/acetaminophen 5/500mg TID or the most appropriate formulary alternative). Participant can also receive up to 2 PRN administrations at the same dose levels as listed above, but not to exceed 2.5g of acetaminophen.
Arm/Group | Experimental: A1 | Placebo Comparator: A2
Number analyzed (Participants) | 8 | 8
units on a scale | 2.20 (1.21) | 2.56 (1.41)

2. Secondary Outcome: Pain Assessment in Advanced Dementia (PAINAD)
Description: Pain intensity observational assessment for persons with severe dementia. Higher scores indicate more pain/discomfort.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Phase B: Open Label: Those participants for whom the study medication was tolerated during Phase A (i.e., the closed label, double-blind phase of the trial) entered a six-week open-label phase.
Arm/Group | Phase B: Open Label
Number analyzed (Participants) | 8
units on a scale | 1.93 (1.98)

ADVERSE EVENTS:
Arm/Group | ALL STUDY PARTICIPANTS
Serious Adverse Events (participants affected / at risk) | 2/11
Other Adverse Events (participants affected / at risk) | 1/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALL STUDY PARTICIPANTS (N=11)
Death (Blood and lymphatic system disorders) | 1 (1) — Sepsis. Not related to study drug/procedures. This participant was in late stages of dementia, at end of life.
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Determined 'related to study drug/procedures' because respiratory distress is a known side effect of the study drug. Participant thus exited from study. This participant was in late stages of dementia.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALL STUDY PARTICIPANTS (N=11)
Serum C02 level dropped (Respiratory, thoracic and mediastinal disorders) | 1 (1) — At regularly scheduled laboratory blood draw, serum C02 level was dropped. Administration of study medication was halted while subject evaluated. C02 level re-evaluated by 2 follow-up lab tests and review by attending physician.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes